CLINICAL TRIAL: NCT03374098
Title: Leland Medical Clinic Patient-Centered Medical Chronic Disease Home Visitation Pilot
Brief Title: Pilot of Home Visitation Services for Patients With a Diabetes Diagnosis
Acronym: LMC-PCMH-H
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Delta Health Alliance (Other)
Collaborators: University of Tennessee (Other); Emory University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 17-036
Record Dates: First submitted 2017-09-14; First posted 2017-12-15 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Diabetes
Keywords: Medicaid; Mississippi
MeSH Terms: conditions — Diabetes Mellitus | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education (Experimental): Attend an hour-long classes once per week for three weeks
  Interventions: Behavioral: Education
- Home Visitation (Experimental): Receive home visits that focus on the social determinants of health and attend hour-long classes once per week for three weeks
  Interventions: Behavioral: Home Visitiation; Behavioral: Education

INTERVENTIONS:
Behavioral: Home Visitiation — The home visit component of the intervention will involve a visit to participants' homes by a social worker, who will assist patients dealing with other health and social problems. Participants will be followed for a minimum of 10 weeks, and additional follow-up visits will be at the discretion of the social worker. They will work with community partners and refer patients when appropriate.
  Community partners could include: Domestic violence services, employment placement, benefit enrollment, community action agency (bill pay, utilities), ACA enrollment, homeless shelter, housing authority, re-housing program
  Arms: Home Visitation
Behavioral: Education — The education component of the intervention will include attending a class once per week for 3 weeks. Classes will be led by a dietician, and may also involve other members of an interdisciplinary team including nurse practitioners, health educators, and community members. Education sessions will be held at 5:30pm on Mondays or Tuesdays, and participants will be provided with a meal. Topics will include:
  * Week 1 (5:30-6:30pm): Importance of self-management of disease, glucometer testing for blood sugars and using home blood pressure monitors, diabetes medication review
  * Week 2 (5:30-7:00pm): Diabetes and Healthy Eating and Exercise - carbohydrate counting, portion control, lifestyle activity, and exercise demonstration activity
  * Week 3 (5:30-6:30pm): Grocery shopping guidelines, label reading, hands on cooking demo

SUMMARY:
This pilot program will assess whether an enhanced PCMH model with more intensive management and intervention can improve chronic disease patient outcomes, improve healthcare delivery, and reduce healthcare costs. Participants in this program are current patients at Leland Medical Clinic and are either enrolled, or eligible to enroll, in Mississippi's Medicaid program. This pilot program will test the effectiveness of high-quality interventions comprising of: (1) an educational intervention focusing on chronic disease management and (2) home visits by a trained community outreach worker.

This pilot program will evaluate both process measures and outcome measures. Examples of process measures include, but are not limited to, the number of patients enrolled in each intervention group, the number of educational classes attended by a unique patient, and the number of home visits a unique patient receives. Examples of outcomes measures include, but are not limited to, change in patient HbA1C levels, change in patient LDL/HDL levels, change in patient blood pressure (systolic and diastolic) levels, and a comparison of patient cost data (total expenditure, expenditures by other major categories like hospital, pharmacy, etc.) After baseline measurements, patient clinical values will be acquired every 3 months for the duration of their engagement.

This pilot project has three specific goals:

Goal 1: Improve healthcare delivery for chronic disease patients enrolled in Mississippi Medicaid.

Goal 2: Improve clinical outcomes for chronic disease patients enrolled in Mississippi Medicaid.

Goal 3: Reduce Mississippi Medicaid costs for chronic disease patients enrolled in this pilot program.

DETAILED DESCRIPTION:
Research Protocol including:

Research procedures:

The aim of this research project is to test whether an enhanced PCMH model with more intensive management and intervention can improve patient outcomes and reduce costs related to chronic disease conditions.

Project eligibility:

* Leland Medical Clinic patient
* Ages 18+
* Medicaid beneficiaries or are Medicaid eligible
* Diagnosis of diabetes and at least one other chronic condition, and an A1c value of 7.5 or above

Leland Medical Clinic patient records will be reviewed to identify potentially eligible patients and a flag will be put on their record for them to be approached at their next office visit for screening, or they could be actively contacted by the clinic by mail or phone.

Once identified as meeting inclusion criteria, patients will be randomized into two additive intervention groups:

1. Education
2. Education + Home Visits

The interventions are additive because if a patient is randomized into group 1, the patient will receive clinical care plus the educational intervention. Meanwhile, if a patient is randomized into group 2, the patient will receive clinical care, education and home visitation. All patients will receive the same level of clinical care regardless of which intervention group patients are randomly assigned.

The first intervention category is an educational program which will be a 10-week series of classes with patients meeting once per week. Led by an interdisciplinary team, including dietitians, nurses, health educators, and community members. Topics of this intervention will include disease self-management support, healthy eating, cooking, exercise, and mental health.

The second intervention category is comprised of education and home visits. A trained community health worker will conduct home visits to assist patients with social, economic and behavioral problems by referring patients, where appropriate, to: domestic violence services, employment placement, benefit enrollment, community action agencies (bill pay, utilities), ACA enrollment, homeless shelters, and housing authorities.

Each patient's clinical outcomes will be measured at the Leland Medical Clinic during regular visits. For example, diabetes patients' HbA1C, LDL/HDL, systolic and diastolic blood pressure, and BMI levels will be recorded every 3 months. Patient satisfaction will also be recorded assessed using the SF-12 patient satisfaction survey, which will be administered every clinical visit.

The subject population will comprise of Leland Medical Clinic's:

1. Diabetes patients, age 18+ with an A1c of 7.5 or above who are enrolled in Mississippi Medicaid; and
2. Diabetes patients, age 18+ with an A1c of 7.5 or above who are eligible for Mississippi Medicaid enrollment.

Recruitment procedures:

Leland Medical Clinic's electronic patient records will be reviewed to identify potentially eligible patients. Potentially eligible patients will be contacted by a study staff member, who will confirm eligibility, consent, and randomize them to one of three intervention groups.

•Length of research procedure and time commitment required of subjects:

The length of this pilot program will be approximately two years. The time length will largely depend upon the speed of recruitment (identifying, consenting, and randomizing). The time commitment required of patients will depend on which intervention group(s) a patient may be enrolled.

If a patient is randomized to the education-only intervention group, a patient will meet for 10 weeks for once per week.

If a patient is randomized to the education plus home visitation intervention group, the patient will meet for the time commitments required for the education intervention (10 weeks for once per week) and participate in at least 10 weeks of home visits (the actual number of required home visits will depend on the needs of the patient).

Location of the study:

The study will primarily take place in Leland Medical Clinic regardless of intervention group. For patients enrolled in the home visitation intervention group, part of the intervention could occur within patients' homes or agreed upon locations.

Methodology:

Based on the results of a power analysis, a minimum of 90 patients or 45 per intervention group will be randomly assigned to an intervention group. Using patient clinical data, patient outcomes will be assessed every 3 months for a total of a year after a baseline measurement which will occur after group randomization.

To statistically analyze these outcomes, differences-in-differences regression models will be performed with HbA1c, cholesterol levels (HDL/LDL), blood pressure levels (systolic, diastolic), and patient Body-Mass Index (BMI) as the outcome variables and using patient age, gender, race, and ethnicity as control variables.

Description of who will gather the data and how they are/will be trained:

Leland Medical Clinic will employ a dietitian and at least one home visitation community health worker. The dietitian and community health worker will collect individual patient process measures covering data pertinent to health education classes and the number of home visits.

Clinical measurements, such as HbA1c, will be collected by clinic staff at Leland Medical Clinic.

Sources of funding:

Funding for this project is awarded annually by the Mississippi Division of Medicaid as approved by the Mississippi State Legislature.

Benefits to the subject or to others:

Leland Medical Clinic patients will benefit from this pilot program through enrollment in high-quality health interventions for managing chronic diseases. Patients living with chronic diseases will have an increased likelihood to receive chronic disease self-management education and case management. Patients will have an increased likelihood to be treated earlier and with appropriate care, which will improve patient health.

Risks -

• Describe the possible risks, discomforts, and inconvenience to the subjects and the precautions that will be taken to minimize them (include physical, psychological and social risks).

There are minimal physical, psychological, or social risks to the subjects.

• Describe appropriate controls, screenings methods, follow-up procedures.

Leland Medical Clinic has installed data security protocols which includes controlling data access and password security. Leland Medical Clinic staff have completed background checks on all project team members. Project team were also trained in HIPAA procedures and compliance. This training will be repeated during the first quarter of each calendar year.

• Describe what constitutes termination from the study before its completion.

Subjects may be terminated from the study if:

1. They die prior to the study's completion;
2. Their participation causes a concern of a threat of physical or psychological threat to themselves, other study subjects, and/or study team members;
3. They choose to opt-out of the study.

   * Describe how confidentiality will be maintained including confidentiality of data collection and who will have access to the data.

Leland Medical Clinic staff members and associated research members complete HIPAA/Privacy training annually. The clinic executes Confidentiality Agreements with its employees and has established controls regarding the use of Protected Health Information (PHI) maintained within all Information Systems which includes:

* Disallowing the disclosure of information/PHI to unauthorized persons without the appropriate consent of the information/PHI owner except as permitted under applicable DHA policy and/or Federal or State law;
* Limiting access to the information/PHI contained in, or obtained from, Information Systems to authorized users;
* Protect Information/PHI against accidental or unauthorized access, modifications, disclosures, or destruction through unauthorized access to any passwords, user identifications, or other information that may be used to access Information Systems, whether those systems belong to DHA or to private parties.

Additionally, Leland Medical Clinic and DHA-affiliated researchers are governed by a Data Use Agreement (DUA) with the Mississippi Division of Medicaid. Data is transferred in a HIPAA compliant, secure environment. Access to the data is limited to health care professionals who have a relationship with the subjects, members of Leland Medical Clinic's project team and the project evaluators.

Informed Consent

Consent is not required as HIPAA permits disclosure as long as Leland Medical Clinic and DHA-affiliated researchers will be sharing patient data with only those health care professionals that also have a relationship with the individual who is the subject of the PHI. Further, the MS Medicaid Notice of Privacy Practices and the application form for Medicaid and CHIP authorize providers to share information with each other. Thus, the DHA can use an "opt out" approach to consent. HIPAA section 164.5220 allows us to share data unless the Medicaid beneficiary asks and the clinic agrees to stop sharing information.

Although not required for this project as explained above, upon initial engagement, patients will be provided an enrollment form to review and sign. This form will explain to patients what is required of them and patients will be advised of how they may opt out of the program.

ELIGIBILITY:
Inclusion Criteria:

* Leland Medical Clinic (LMC) patients
* Medicaid beneficiary or no insurance
* Active diabetes diagnosis
* Diagnosis of at least one other chronic condition (COPD, Hypertension, chronic kidney disease, CHF
* Baseline HbA1c 7.0 or above.

Exclusion Criteria:

- Patients with active psychoses will not be eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in HbA1C values | Six months and three months before enrollment, at enrollment, three and six months follow-ups
  Data recorded in electronic health records system

SECONDARY OUTCOMES:
ED visits | Baseline and six-month follow-up
  Emergency department utilization measured by Medicaid claims data
Changes in LDL values | Six months and three months before enrollment, at enrollment, three and six months follow-ups
  Data recorded in electronic health records system
Changes in blood pressure values | Six months and three months before enrollment, at enrollment, three and six months follow-ups
  Data recorded in electronic health records system
Total medical costs | End of enrollment in intervention and six month follow-up
  Using electronic health records and practice management data along with Medicaid claims data
Medication adherence | At enrollment in intervention, six month follow-up
  Morisky Medication Adherence Scale (0 to 4 scale with higher number demonstrating low adherence)
Patient Engagement and Activation | At enrollment in intervention, six month follow-up
  Patient Activation Measure (22 questions, scored 0 to 100, with higher number demonstrating more patient engagement)
Diet | At enrollment in intervention, six month follow-up
  Rapid Eating Assessment for Patients (27 questions, with higher number demonstrating less healthy eating habits)
Hospitalizations | Baseline and six-month follow-up
  Hospital utilization measured by Medicaid claims data
Physical Activity | At enrollment in intervention, six month follow-up
  Rapid Eating Assessment for Patients (27 questions, with higher number demonstrating less healthy eating habits)

CONTACTS AND LOCATIONS:
Overall Officials: Karen C Matthews, Principal Investigator — Delta Health Alliance
Locations (1):
- Leland Medical Clinic, Leland, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No